CLINICAL TRIAL: NCT03481608
Title: Production of a LRH-1 Ligand in Humans: A Randomized,Controlled, Cross-Over Feeding Trial
Brief Title: The Effect of Dietary Lauric Acid on the Production of the LRH-1 Ligand, Dilauroylphosphatidylcholine
Acronym: DLauricPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1802007735
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Diet Modification
Keywords: fatty acid; nutrition; metabolism; lauric acid; dilauroylphosphatidylcholine; lrh-1
MeSH Terms: interventions — lauric acid; Coconut Oil; Olive Oil

STUDY DESIGN:
Intervention Model Description: Acute feeding study. Participants will arrive at our Human Metabolic Research Unit on 2 separate occasions. Participants will be randomized to consume 1 of 2 shake on each occasion. Shakes will be prepared with 2 tablespoons of either control (olive) or intervention (coconut) oils.
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention oil (single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Oil Shake (Active Comparator): Intervention: No Lauric Acid
  A breakfast shake made from a complete meal shake will be prepared with water and supplemented with 2 tablespoons of olive oil.
  Interventions: Other: No Lauric acid (olive oil)
- Coconut Oil Shake (Experimental): Intervention: Lauric Acid
  A breakfast shake made from a complete meal shake will be prepared with water and supplemented with 2 tablespoons of coconut oil.
  Interventions: Other: Lauric acid (coconut oil)

INTERVENTIONS:
Other: Lauric acid (coconut oil) — A breakfast shake made from a complete meal shake will be prepared with water and supplemented with 2 tablespoons of coconut oil.
  Arms: Coconut Oil Shake
Other: No Lauric acid (olive oil) — A breakfast shake made from a complete meal shake will be prepared with water and supplemented with 2 tablespoons of olive oil.
  Arms: Olive Oil Shake

SUMMARY:
A phosphatidylcholine species enriched with lauric acid at both the sn-1 and sn-2 positions, dilauroylphosphatidylcholine (DLPC), was recently identified as a ligand for the nuclear receptor, liver receptor homolog-1 (LRH-1). To date, DLPC has not been reported in vitro or in vivo, and has yet to be catalogued in the human metabolomics database. This intervention trial aims to determine the impact of consumption of dietary lauric acid, in the form of coconut oil (49% lauric acid), can facilitate the production of DLPC in humans.

DETAILED DESCRIPTION:
A phosphatidylcholine species enriched with lauric acid at both the sn-1 and sn-2 positions, dilauroylphosphatidylcholine (DLPC), was recently identified as a ligand for the nuclear receptor, liver receptor homolog-1 (LRH-1). LRH-1 has notable roles in regulating sterol metabolism, with downstream impacts on reproductive capacity, bile acid production, glucose metabolism, and cell proliferation. Manipulation of LRH-1 activity via ligand-inducing binding and activation has the potential to act as a therapy in certain metabolic disorders, such as type 2 diabetes. To date, the LRH-1 ligand, DLPC, has not been reported in vitro or in vivo, and has yet to be indexed in the Human Metabolomics Database, suggesting that it's therapeutic potential is limited to pharmacological administration. The investigators' forthcoming unpublished research tested the hypothesis that the lack of DLPC in physiological systems results from substrate insufficiency, and have observed that consumption of dietary lauric acid facilitates the production of DLPC in animal models, and addition of lauric acid to the culture media of cells additionally leads to its production. A single acute gavage of coconut oil results in the production of DLPC in the intestine and export in the serum 1-2 hours post-gavage. To extend this work to humans, the investigators are undertaking an acute, randomized, cross-over trial of dietary lauric acid consumption. This intervention trial aims to determine whether dietary lauric acid, in the form of coconut oil (49% lauric acid), can facilitate the production of DLPC in humans. The investigators have hypothesized that consumption of a single breakfast shake containing coconut oil will result in DLPC in post-prandial serum. Participants will be invited to the Cornell University Human Metabolic Research Unit (HMRU) on 2 separate occasions to consume 1 of 2 breakfast shake , delivered in random order. Shakes will be made with either 2 tablespoons of olive oil (control) or coconut oil (intervention). Participants will arrive to the HMRU fasted and provide a baseline blood sample, prior to consumption of the breakfast shake ; at 2, 4, and 6 hours following the meal, participants will provide additional blood samples. Prior to and throughout the duration of the study, participants will be asked to avoid consumption of tropical oils. Lauric acid is typically a minimal component of the common diet, though substantial intakes can occur with the consumption of tropical oils, such as coconut oil or palm kernel oil. Lauric acid is considered one of the three primary hypercholesterolemic saturated fatty acids and is currently not recommended to constitute a major component of the diet; participants for whom a cholesterol lowering diet is recommended will not be able to enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with the study protocol
* Ability to overnight fast
* Willingness to donate blood
* 'generally healthy'

Exclusion Criteria:

* self-reported regular consumption of tropical oils or supplements containing lauric acid
* self-reported food allergies to shake ingredients
* medical conditions where blood draws or fasting may be contraindicated
* major gastrointestinal conditions, such as inflammatory bowel disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
DLPC in Postprandial Serum | 6 hours postprandial
  The presence of DLPC in postprandial serum will be measured using Liquid Chromatography Tandem Mass Spectrometry

SECONDARY OUTCOMES:
Serum Total Bile Acids | 6 hours postprandial
  Serum total bile acids may be measured following shake consumption using a colorimetric assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Metabolic Research Unit, Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data, including mass spectra, can be made available upon request.